CLINICAL TRIAL: NCT07383389
Title: Validation of the Turkish Respiratory Distress Observation Scale Using End-Tidal Carbon Dioxide in Critical Care Patients
Brief Title: Validation of the Turkish RDOS Using End-Tidal Carbon Dioxide
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yunus Emre Tutuneken, Assistant Professor, Istinye University
Other Study IDs: 115
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Critical Care, Intensive Care; Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critical illness patients

SUMMARY:
Dyspnea is a complex and distressing symptom frequently observed in critically ill patients and is associated with increased morbidity, mortality, and prolonged intensive care unit (ICU) stay. Although dyspnea is inherently subjective, accurate assessment of its presence and severity is essential for appropriate clinical decision-making and treatment planning. In routine clinical practice, dyspnea is commonly assessed using patient self-report scales; however, this approach is not feasible in patients who are unable to communicate due to impaired consciousness, cognitive dysfunction, mechanical ventilation, sedation, or severe illness. Consequently, there is a critical need for valid and reliable observational tools that allow healthcare professionals to assess respiratory distress in non-communicative patients.

The Respiratory Distress Observation Scale (RDOS) is an eight-item observational instrument originally developed to assess respiratory distress in patients who cannot self-report dyspnea. The scale evaluates observable physiological and behavioral indicators, including respiratory rate, heart rate, use of accessory muscles, paradoxical breathing, nasal flaring, grunting, restlessness, and facial expression. RDOS has demonstrated acceptable reliability and validity in various patient populations and has been translated into multiple languages. A Turkish version of the RDOS has recently undergone linguistic and cultural adaptation; however, its validity has not yet been examined using an objective physiological reference standard.

End-tidal carbon dioxide (ETCO₂), measured via capnography, provides a continuous, non-invasive indicator of ventilatory status and has been widely used in critically ill patients to monitor ventilation and respiratory adequacy. Alterations in ETCO₂ values may reflect changes in respiratory mechanics, ventilation-perfusion mismatch, and respiratory distress. Therefore, ETCO₂ represents a clinically relevant objective parameter for examining the concurrent validity of observational dyspnea assessment tools.

The primary objective of this study is to evaluate the validity of the Turkish version of the Respiratory Distress Observation Scale by examining its relationship with end-tidal carbon dioxide levels in critically ill adult patients hospitalized in the intensive care unit. This prospective observational study will be conducted over a six-month period in the ICU of a tertiary care hospital. A total of 64 adult patients aged 18 to 85 years who experience dyspnea and meet the inclusion criteria will be enrolled. Patients who are fully dependent on mechanical ventilation or have severe central nervous system disorders affecting respiratory control will be excluded.

Following ethical approval and informed consent obtained from patients' legal representatives, demographic and clinical data will be collected from medical records. Physiological parameters including oxygen saturation, respiratory rate, heart rate, blood pressure, body temperature, arterial blood gas values, and ETCO₂ will be recorded simultaneously. Disease severity will be assessed using the Acute Physiology and Chronic Health Evaluation II (APACHE II) score. The Turkish RDOS will be administered by a trained evaluator, and capnography measurements will be performed concurrently using appropriate mainstream or sidestream techniques depending on the patient's airway status.

Statistical analyses will include descriptive statistics and correlation analyses to examine the relationship between RDOS scores and ETCO₂ values. Concurrent and convergent validity will be evaluated using Pearson or Spearman correlation coefficients, depending on data distribution. It is hypothesized that higher RDOS scores, indicating more severe respiratory distress, will be associated with altered ETCO₂ levels, supporting the validity of the Turkish RDOS as an objective observational measure of dyspnea in critically ill patients.

The findings of this study are expected to provide important evidence supporting the clinical utility of the Turkish version of the Respiratory Distress Observation Scale for assessing respiratory distress in patients who are unable to self-report dyspnea. Establishing its validity against an objective physiological marker may facilitate more accurate monitoring of dyspnea, improve symptom management, and enhance the quality of care in intensive care settings.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Having a diagnosis of lung or pleural cancer, chronic kidney failure, congestive heart failure, COPD, asthma, or pneumonia presenting with dyspnea,
* Being specifically referred for treatment of dyspnea,
* Having been in the intensive care unit for at least one day,
* Participation in the study must be consented to by the individual or a family member.

Exclusion Criteria:

* Being completely ventilator-dependent,
* Having a diagnosis of central nervous system disease (quadriplegia, bulbar ALS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 85 years who are hospitalized in the intensive care unit with clinically diagnosed dyspnea and underlying cardiopulmonary or systemic conditions. Eligible participants are patients who are unable to reliably self-report respiratory distress due to critical illness or impaired communication. Patients who are fully dependent on mechanical ventilation or have severe central nervous system disorders affecting respiratory control are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The concurrent validity of the Turkish version of the Respiratory Distress Observation Scale (RDOS) | 4 Months
  The concurrent validity of the Turkish version of the Respiratory Distress Observation Scale (RDOS), assessed by examining the relationship between RDOS total scores and end-tidal carbon dioxide (ETCO₂) levels in critically ill patients. The strength and direction of the association between RDOS scores and ETCO₂ values measured simultaneously via capnography will be analyzed to determine whether the RDOS reflects objective ventilatory status in patients unable to self-report dyspnea.